CLINICAL TRIAL: NCT04498065
Title: MYocardial DOmmages Related to COVID-19
Acronym: DOMY COVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: COTTIN AOIc 2020
Record Dates: First submitted 2020-08-03; First posted 2020-08-04 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Covid19; Non Ischemic Myocardial Injury; Myocardial Infarction; Myocarditis; Troponin Elevation
MeSH Terms: conditions — COVID-19; Myocardial Infarction; Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: COVID positive and Troponin positive
  Interventions: Biological: Biological data; Other: Clinical data
- B: COVID positive and Troponin negative
  Interventions: Biological: Biological data; Other: Clinical data

INTERVENTIONS:
Biological: Biological data — Biological data
Other: Clinical data — Clinical data

SUMMARY:
Myocardial injury, as assessed by elevation of cardiac troponins (Tnc), is frequent among patients with COVID-19. Although rare autopsy cases reported COVID-19 related myocardial inflammation, the origin of Tnc elevation is unknown to date. Several cardiac causes, such as myocarditis, non-ischemic myocardial injury (NIMI), or myocardial infarction (MI) may lead to Tnc kinetic. Our work will test the hypothesis that during SARS-Cov2 infection, the elevation of cardiac biomarkers could be linked to the occurrence of myocarditis.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive patient hospitalized < 72 h after symptoms onset with troponin assessement.

Exclusion Criteria:

* patients hospitalized > 72h after symptom onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to CHU Dijon Bourgogne for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
characterize the myocardial damage associated with CoV-2 SARS infection | Through study completion, an average of 2 years
  Myocardtitis diagnosis in patients COVID+ and troponin+

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France